CLINICAL TRIAL: NCT05455723
Title: Tracheal Tube Cuff Inflation-Deflation Method for Video Assisted Laryngoscope Nasal Intubation in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Aiman Al-Touny, Lecturer of Anesthesia and Intensive Care, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4523#
Record Dates: First submitted 2022-07-10; First posted 2022-07-13 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Airway Management; Nasal Intubation; Video Laryngoscope
Keywords: Magill forceps; Inflation-deflation technique; Video-assisted Laryngoscope; Nasal intubation

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The nasal intubation will be performed behind an opaque screen so that observer could not see which approach will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inflation-Deflation Group (Active Comparator): Group A (45 patients): Phase 2 of ETT intubation will be performed with tracheal tube cuff inflation-deflation method. Tracheal tube cuff will be inflated with 15-20 ml of air (volume of air is depending on the level of larynx). Once the tip of ETT at the laryngeal inlet, the cuff of ETT will be deflated and advanced into the trachea.
  Interventions: Procedure: Inflation-deflation technique
- Magill Forceps Group (Active Comparator): Group B (45 patients): Phase 2 of ETT intubation will be performed using the Magill forceps to guide the ETT tip to pass through the pharynx and glottis into the trachea.
  Interventions: Procedure: Magill forceps technique

INTERVENTIONS:
Procedure: Inflation-deflation technique — Inflation-Deflation Technique: The tracheal tube cuff will be inflated with 15-20 ml of air (volume of air is depending on the level of larynx). Once the tip of ETT at the laryngeal inlet, the cuff of ETT will be deflated and advanced into the trachea.
  Arms: Inflation-Deflation Group
Procedure: Magill forceps technique — The Magill forceps to guide the ETT tip to pass through the pharynx and glottis into the trachea.
  Arms: Magill Forceps Group

SUMMARY:
The goal of this clinical trial is to compare cuff inflation deflation method versus conventional method using Magill forceps in adult patients scheduled for elective surgery dental or maxillofacial that need nasal intubation. The study question:

Is cuff inflation deflation method for nasal intubation takes a short time than the conventional method using Magill forceps in adult patients scheduled for elective surgery dental or maxillofacial?

We will compare the inflation deflation technique with the Magill forceps technique for nasal intubation in adult patients to see if the inflation deflation technique will take less time and associated with less side effects like cuff perforation and mucosal injury.

Participants will [describe the main tasks participants will be asked to do, interventions they'll be given and use bullets if it is more than 2 items].

DETAILED DESCRIPTION:
Magill forceps is used to maneuver the endotracheal tube (ETT) in the posterior oropharynx and place its tip into the laryngeal inlet. While the Magill forceps are useful in guiding the nasotracheal tube past the vocal cords, care must be taken to avoid excessive maneuvering in order to minimize the risk of local trauma and rupture of the nasotracheal tube balloon.

Cuff inflation-deflation method can reduce the apnea time in the adult patients. This, in turn, could point to a reduction in the complications (as desaturation and cardiac arrhythmia) that associated with the prolonged-time procedure.

Written informed consent will be obtained from all patients participating in the trial. The trial will be registered prior to patient enrollment. Ninety patients between the ages of 18 and 60 years with American Society of Anesthesiologists (ASA) physical status I -II , scheduled for elective surgery (dental and maxillofacial) will be enrolled in a prospective randomized observer blinded clinical trial. Patients, who have coagulopathies, have upper airway abnormalities, at risk for aspiration or patient's refusal will be excluded from the study.

Materials and methods

Airway management is subdivided into phases:

Phase 1 :Passage of the endotracheal tube through the nose into the pharynx Phase 2 : Video-laryngoscope-guided passage of the endotracheal tube through the pharynx into the trachea.

Patients will be randomized into 2 groups according to phase 2:

Group A (45 patients) will be performed with tracheal tube cuff inflation-deflation method. Tracheal tube cuff will be inflated with 15-20 ml of air (volume of air is depending on the level of larynx). Once the tip of ETT at the laryngeal inlet, the cuff of ETT will be deflated and advanced into the trachea.

Group 2 (45 patients) will be performed using the Magill forceps to guide the ETT tip to pass through the pharynx and glottis into the trachea.

Patients will be randomly assigned on a one-to-one ratio. Randomization will be performed outside the study center by means of a computer generated random- numbers table. Group allocation will be concealed in sealed opaque envelopes that will not be opened till the last practical moment.

The nasal intubation will be performed behind an opaque screen so that observer could not see which approach will be used. All procedures were performed preoperatively by the attending anesthetists, who have the same substantial expertise (at least 3 years) in the video laryngoscopy assisted nasal intubation in adult patients. Patient demographics, type and duration of surgery, and the patient's ASA physical status will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-III
* Scheduled for elective surgery (dental and maxillofacial) in need for nasal intubation.

Exclusion Criteria:

* Patients, who have coagulopathies,
* Have upper airway abnormalities,
* At risk for aspiration or by reasons of
* Parent's refusal will be excluded from the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2025-02-25 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
The time period for the second phase of nasal intubation | Intraoperaotive
  The time in seconds for the second phase nasal intubation(from the tip of endotracheal tube will be placed in pharynx till it pass the vocal cords

SECONDARY OUTCOMES:
to test whether the inflation-deflation method would decrease the need for Magill forceps in video laryngoscopy assisted nasal intubation in pediatric patients compared with the conventional non-cuff inflation approach. | Intraoperaotive
  The percentage of patients who did not require Magill forceps for nasal intubation success was recorded.
The number of attempts required for successful nasal intubation. | Intraoperaotive
  number of trials, how many numbers of attempts the investigator take for successful nasal intubation
Amount of injected air for cuff inflation | Intraoperaotive
  Amount of injected air in ml, how many air injected in the cuff balloon to make the tip of endotracheal tube advanced into the trachea
Assessment of side effects of using Magill forceps during nasal intubation | Intraoperaotive
  A 4-point scale: 1- No epistaxis; 2-Mild epistaxis (blood on the tracheal tube only); 3- Moderate epistaxis (blood pooling in the pharynx); 4- Severe epistaxis (blood in the pharynx sufficient to impede intubation)
Evaluation of oxygenation state during nasal intubation | preoperative and intraoperative
  rate of oxygen drop during the procedure
evaluate the anesthetists' experience of using the inflation-deflation method for nasal intubation. | 20 minutes after patient recovery
  score 1 to 5 A five-point Likert scales for: How likely is it that anesthetist would recommend the same used inflation-deflation method to practice a colleague in the future (not at all/ slightly/ moderately/ very/ extremely: where 1 is not at all, 3 is moderate,5 is extremely
Need for external compression and need for help | Intraoperaotive
  Need for external tracheal compression and need for help
need of endotracheal tube rotation | Intraoperaotive
  need of endotracheal tube rotation and the degree of rotation 90, 180 0r 360 degree

CONTACTS AND LOCATIONS:
Overall Officials: Tarek F. Tammam, Professor, Principal Investigator — Suez Canal University
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No